CLINICAL TRIAL: NCT05074875
Title: Post COVID-19 Hypoxemic Respiratory Failure Residual Pathophysiologic Outcomes
Brief Title: COVID-19 Respiratory Outcomes Registry
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 20-05022161
Record Dates: First submitted 2021-04-06; First posted 2021-10-12 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires; Patient Reported Outcome Measures; Blood Specimen Collection; Biomarkers; Physical Examination; Vital Signs; Hand Strength; Spirometry; Walk Test; Sequence Tagged Sites

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, and RNA will be collected at baseline, week 4, week 24, week 36, and week 48 to identify biomarkers that may put patients with COVID-19 at greater risk for development and/or progression of chronic fibrotic interstitial lung disease (ILD). Blood for DNA will be collected at baseline to assess whether genetic factors may increase the risk for development and/or progression of chronic fibrotic interstitial lung disease (ILD).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1: Subjects with a diagnosis of hypoxemic respiratory failure associated with COVID-19 who meet the inclusion and exclusion criteria will be eligible for participation in this study.
  Cohort 1 subjects will undergo Visit 0 after informed consent is obtained. Eligible subjects will return for follow-up at Visits 2, 3, and 4, at weeks 24, 36, and 48 weeks
  Interventions: Other: Questionnaires and Patient Reported Outcomes (PROs); Diagnostic Test: Nasal Swab COVID-19 reverse transcription polymerase chain reaction test (RT-PCR); Genetic: Blood Samples for Biomarkers; Diagnostic Test: High Resolution Computed Tomography; Diagnostic Test: Physical Exam and Vital Signs; Diagnostic Test: Medical Research Council Sum Score; Diagnostic Test: Hand Grip Strength; Diagnostic Test: Spirometry; Diagnostic Test: Diffusing Capacity of Carbon Monoxide; Diagnostic Test: 6 Minute Walk Test; Diagnostic Test: Sit to Stand (STS) Measurement
- Cohort 2: Subjects with a diagnosis of hypoxemic respiratory failure associated with COVID-19 who meet the inclusion and exclusion criteria will be eligible for participation in this study.
  Cohort 2 subjects will undergo Visit 1, within 4 (+/- 2) weeks of hospital discharge or outpatient infection, after informed consent is obtained. Eligible subjects will return for follow-up Visits 2, 3, and 4, at weeks 24, 36, and 48 weeks.
  Interventions: Other: Questionnaires and Patient Reported Outcomes (PROs); Diagnostic Test: Nasal Swab COVID-19 reverse transcription polymerase chain reaction test (RT-PCR); Genetic: Blood Samples for Biomarkers; Diagnostic Test: High Resolution Computed Tomography; Diagnostic Test: Physical Exam and Vital Signs; Diagnostic Test: Medical Research Council Sum Score; Diagnostic Test: Hand Grip Strength; Diagnostic Test: Spirometry; Diagnostic Test: Diffusing Capacity of Carbon Monoxide; Diagnostic Test: 6 Minute Walk Test; Diagnostic Test: Sit to Stand (STS) Measurement
- Cohort 3a: Subjects with a diagnosis of hypoxemic respiratory failure associated with COVID-19 who meet the inclusion and exclusion criteria will be eligible for participation in this study.
  Cohorts 3a and 3b subjects will undergo their first study visit between 6 and 24 weeks of hospital discharge or outpatient infection, after informed consent is obtained. Participants should not be scheduled for chest HRCTs less than 12 weeks apart, however all subjects should have an HRCT done at Week 24 for analysis purposes. To prevent scheduling of HRCTs within less than 12 weeks.
  Subjects enrolled within ≤ 12 weeks of hospital discharge or outpatient COVID- 19 infection will undergo their first study visit at Visit 1 (Weeks 6-12).
  Interventions: Other: Questionnaires and Patient Reported Outcomes (PROs); Diagnostic Test: Nasal Swab COVID-19 reverse transcription polymerase chain reaction test (RT-PCR); Genetic: Blood Samples for Biomarkers; Diagnostic Test: High Resolution Computed Tomography; Diagnostic Test: Physical Exam and Vital Signs; Diagnostic Test: Medical Research Council Sum Score; Diagnostic Test: Hand Grip Strength; Diagnostic Test: Spirometry; Diagnostic Test: Diffusing Capacity of Carbon Monoxide; Diagnostic Test: 6 Minute Walk Test; Diagnostic Test: Sit to Stand (STS) Measurement
- Cohort 3b: Subjects with a diagnosis of hypoxemic respiratory failure associated with COVID-19 who meet the inclusion and exclusion criteria will be eligible for participation in this study.
  Cohorts 3a and 3b subjects will undergo their first study visit between 6 and 24 weeks of hospital discharge or outpatient infection, after informed consent is obtained. Participants should not be scheduled for chest HRCTs less than 12 weeks apart, however all subjects should have an HRCT done at Week 24 for analysis purposes. To prevent scheduling of HRCTs within less than 12 weeks.
  Subjects enrolled ≥ 12 weeks from hospital discharge or outpatient COVID- 19 infection will undergo their first visit within 4 weeks before week 24. Subjects that are enrolled into Cohort 3 will be followed until Week 72.
  Interventions: Other: Questionnaires and Patient Reported Outcomes (PROs); Diagnostic Test: Nasal Swab COVID-19 reverse transcription polymerase chain reaction test (RT-PCR); Genetic: Blood Samples for Biomarkers; Diagnostic Test: High Resolution Computed Tomography; Diagnostic Test: Physical Exam and Vital Signs; Diagnostic Test: Medical Research Council Sum Score; Diagnostic Test: Hand Grip Strength; Diagnostic Test: Spirometry; Diagnostic Test: Diffusing Capacity of Carbon Monoxide; Diagnostic Test: 6 Minute Walk Test; Diagnostic Test: Sit to Stand (STS) Measurement

INTERVENTIONS:
Other: Questionnaires and Patient Reported Outcomes (PROs) — * EuroQol 5 Dimensional Quality of Life Questionnaire (EQ-5D).
  * St. George's Respiratory Questionnaire (SGRQ)
  * Impact of Events Scale Revised (IES-R)
  * Generalized Anxiety Disorder 7-Item (GAD-7)
  * Patient Health Questionnaire (PHQ-9)
Diagnostic Test: Nasal Swab COVID-19 reverse transcription polymerase chain reaction test (RT-PCR) — If required by the local site's COVID-19 guidelines, subjects should have the COVID-19 RT-PCR Nasal Swab collected at the beginning of the visit or within 5 days prior to the scheduled visit.
Genetic: Blood Samples for Biomarkers — Venous blood will be collected using pre-labeled tubes.
Diagnostic Test: High Resolution Computed Tomography — Subjects will have HRCTs at Visits 1, 2, 3, and 4. Inpatient HRCT scans will be collected during the baseline visit (V0 or V1)
Diagnostic Test: Physical Exam and Vital Signs — A complete physical exam, including height, weight, general appearance, neck, lungs, cardiovascular system, abdomen, extremities, and skin will be performed at Visit 1.A brief physical exam will be completed at subsequent visits, including weight, general appearance, lungs, cardiovascular symptoms, extremities, and other body systems pertinent to the participants health status, at the discretion of the investigator.
  Blood pressure, heart rate, and oxygen saturation will be collected at all visits, prior to blood draws and after subjects have rested.
Diagnostic Test: Medical Research Council Sum Score — The Medical Research Council Sum Score (MRC-SS) is used globally to detect peripheral muscle strength and to help diagnose ICU-acquired muscle weakness. The MRC-SS ranging from 0 (complete paralysis) to 60 (normal).
Diagnostic Test: Hand Grip Strength — Each subject will have hand grip strength measured at each visit. This is being done in order to assess the maximum isometric strength of hand and forearm muscles.
Diagnostic Test: Spirometry — Spirometry will be assessed at Visits 1, 2, 3 and 4. Each site will use its own spirometry machine. Each subject should use the same machine at each visit and conduct measurements at approximately the same time. Before any testing, the maneuver should be demonstrated to the subject. The spirometry should be reviewed by the investigator.
Diagnostic Test: Diffusing Capacity of Carbon Monoxide — The site will use its own DLCO equipment for measurements at Visits, 1, 2, 3, and 4. The Single-breath DLCO maneuver will be carried out in accordance with the 2017 American Thoracic Society/European Respiratory Society (ATS/ERS) guidelines. Subjects should use the same device at approximately that same time at each visit. The maneuver should be demonstrated to the subject prior to the test.
Diagnostic Test: 6 Minute Walk Test — The 6 Minute Walk Test (6MWT) will assess exercise capacity and tolerance. 6MWTs will be conducted at Visits 1, 2, 3, and 4.
  The procedure of the 6MWT should be explained and demonstrated to the subject prior to the start of the test.
Diagnostic Test: Sit to Stand (STS) Measurement — The STS will be conducted at Visits 1, 2, 3, and 4 to assess the physical functioning of the adult participants.

SUMMARY:
This is a 48-week, observational study looking to see if the inflammatory process of hypoxemic respiratory failure associated with COVID-19 leads to progressive pulmonary fibrosis. Inpatient, as well as outpatient adults with recent COVID-19 hospitalization will be recruited. Data from hospitalization will be collected and subjects will return to the center for follow-up visits. Subjects will undergo the following procedures: High Resolution Computed Tomography (HRCT) of the chest, Pulmonary Function Tests (PFT), Muscle Strength Measurement, and blood draw for biomolecular data such as biomarkers found in ribonucleic acid (RNA), deoxyribonucleic acid (DNA), serum, and plasma. Quality of Life (QoL) measurements will also be collected through the study.

DETAILED DESCRIPTION:
This is a multi-center, observational, and prospective study collecting data on subjects who were hospitalized with hypoxemic respiratory failure associated with COVID-19 or patients who have evidence of an outpatient COVID-19 infection that have been treated with supplemental oxygen.

A total of approximately 300 subjects will be enrolled in the study. Subjects will be enrolled into one of 3 cohorts.

Cohort 1: Inpatient Enrollment: Subjects enrolled while hospitalized for COVID-19, prior to discharge.

Cohort 2: Outpatient Enrollment: Subjects enrolled up to 4 weeks after discharge from hospitalization for COVID-19 or 4 weeks post their outpatient COVID -19 infection.

Cohort 3: Outpatient Enrollment: Subjects enrolled between 6 and 24 weeks after discharge from hospitalization for COVID-19 or 6 and 24 weeks post their outpatient COVID -19 infection. Cohort 3 will be sub-divided into 3a and 3b depending on the timepoint of enrollment.

After signing the Informed Consent Form, the screening visit will be performed. Screening and enrollment can occur at Visit 0 (inpatient) or Visit 1 (outpatient). Following completion of Visit 0 or 1 the subjects' data will be assessed by the investigator to confirm eligibility and a decision will be made if the patient is to be enrolled. If not the reason for non-enrollment will be listed in the trial log.

Each subject will either have a total of 4 or 5 visits, depending on if subjects complete enrollment while still admitted to the hospital (Visit 0) or at Visit 1. At weeks 4, 24, 36, 48, all subjects will complete questionnaires, have physical exams, spirometry test with DLCO, HRCTs, 6MWTs, blood draws, and review of medical history since the previous visit.

The primary analysis of this study will be performed once the last enrolled subject reaches Week 48. At that time, there will be a data-base lock. Unless otherwise noted, Visit 1 is treated as baseline measurement. In addition, for patients enrolled at discharge, a second set of analysis will be performed treating Visit 0 as baseline for the measurements collected at Visit 0.

Aim 1: To identify whether the trajectory of COVID-19 associated respiratory failure results in progressive pulmonary fibrosis with clinical features or biomolecular changes.

Aim 2: To identify biomarkers that may indicate those patients at risk for developing a chronic fibrotic HRCT pattern that may go on to progression.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent consistent with International Conference on Harmonization Tripartite Guideline for Good Clinical Practice (ICH-GCP) and local laws signed prior to entry into the study
2. Male or female ≥ 18 years of age at the time of consent
3. SARS-CoV-2 positive confirmed by a positive serology or PCR or antigen test
4. COVID-19 induced hypoxemia or reduced oxygen saturation requiring treatment with supplemental oxygen.
5. COVID-19 hospital discharge date or outpatient COVID-19 infection within 24 weeks of enrollment

Exclusion Criteria:

1. Diagnosed with Fibrotic Interstitial Lung Disease (ILD) prior to COVID-19 infection.
2. Prior treatment with an antifibrotic agent, including nintedanib or pirfenidone
3. Pregnant women or women planning on becoming pregnant in the next 12 months
4. Patients planned for discharge from the hospital to hospice
5. Patients with significant cognitive impairment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with a diagnosis of COVID-19 who require therapy with supplemental oxygen and who meet the inclusion and exclusion criteria will be eligible for participation in this study.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Change in fibrotic and non-fibrotic interstitial opacities on chest HRCT at 48 weeks after hospitalization for COVID-19 or outpatient COVID-19 infections which require treatment with supplemental oxygen | 48 Weeks
  Categorized after exploratory analysis as improved, stable or worsened fibrotic changes seen on chest HRCT.

SECONDARY OUTCOMES:
Changes from baseline and evidence of disease progression seen on high resolution computed tomography | 72 Weeks
  Percentage of subjects with evidence of disease progression by HRCT changes from baseline to 24, 36, 48 and 72 weeks.
Changes from baseline and evidence of disease progression on pulmonary function testing | 72 weeks
  Relative change in Forced Vital Capacity percent predicted (FVC) from baseline to 24, 36, 48 and 72 weeks.
Changes from baseline and evidence of disease progression seen on pulmonary function testing | 72 weeks
  Relative change in Diffusing Capacity of Carbon Monoxide percent predicted (DLCO) from baseline to 24, 36, 48 and 72 weeks.
Changes from baseline and evidence of disease progression see on pulmonary function testing | 72 weeks
  Change in Maximum Inspiratory (PI Max) and Maximum Expiratory (PE Max) [cm H2O] from baseline to 24, 36, 48 and 72 weeks.
Changes from baseline and evidence of disease progression via 6 Minute Walk Test | 72 weeks
  Change from baseline 6 Minute Walk Test (6MWT) distance (feet) from baseline to 24, 36, 48 and 72 weeks.
Change in pre- and post- six minute walk test Borg Scale Dyspnea score from baseline and at 12, 24, and 48 weeks. | 72 weeks
  The top of the scale, "0 or nothing at all," means no breathlessness at all. The bottom of the scale, "10 or maximal," means the most severe breathlessness that you have ever experienced or could imagine experiencing from baseline to 24, 36, 48 and 72 weeks.
Change in pre- and post- six minute walk test Borg Scale Fatigue score from baseline and at 12, 24, and 48 weeks. | 72 weeks
  The top of the scale, "0 or nothing at all," means no fatigue at all. The bottom of the scale, "10 or maximal," means the most severe fatigue that you have ever experienced or could imagine experiencing from baseline to 24, 36, 48 and 72 weeks.
Changes from baseline and evidence of disease progression by Hand Grip Strength | 72 weeks
  Change in Hand Grip Strength value (kg) via hand dynamometer from baseline to 24, 36, 48 and 72 weeks.
Changes from baseline and evidence of disease progression per the Quality of Life reported outcomes. EuroQol-5D (EQ-5D) | 72 weeks
  Change from baseline Quality of Life (QoL) questionnaires from baseline to 24, 36, 48 and 72 weeks.
  EuroQol-5D (EQ-5D) capture health status by asking 5 questions and by using a visual analog scale (0-100)
Changes from baseline and evidence of disease progression per the Quality of Life reported outcomes. St. George's Respiratory Questionnaire (SGRQ) | 72 weeks
  Change from baseline Quality of Life (QoL) questionnaires from baseline to 24, 36, 48 and 72 weeks.
  St. George's Respiratory Questionnaire (SGRQ)
  Patients respond to different prompts by checking off the amount of respiratory symptom occurrences.
  Other prompts require true or false responses.
Changes from baseline and evidence of disease progression per the Quality of Life reported outcomes. Generalized Anxiety 7-Item (GAD-7) | 72 weeks
  Change from baseline Quality of Life (QoL) questionnaires from baseline to 24, 36, 48 and 72 weeks.
  Generalized Anxiety 7-Item (GAD-7) is a 7-item tool used to measure anxiety in patients. Each question is answered on a scale of 0-3
  0- Not at all
  1. Several Days
  2. More than half the days
  3. Nearly every day
  Score indications:
  0-4: minimal anxiety 5-9: mild anxiety 10-14: moderate anxiety 15-21: severe anxiety
Changes from baseline and evidence of disease progression per the Quality of Life reported outcomes. Patient Health Questionnaire 9 (PHQ-9) | 72 weeks
  Change from baseline Quality of Life (QoL) questionnaires from baseline to 24, 36, 48 and 72 weeks.
  Patient Health Questionnaire 9 (PHQ-9)
  This is a 9-item questionnaire. Questions are answered from 0-3
  0- Not at all
  1. Several Days
  2. More than half the days
  3. Nearly every day
Changes from baseline and evidence of disease progression per the Quality of Life reported outcomes- Impact of Events Scale Revised (IES-R) | 72 weeks
  Change from baseline Quality of Life (QoL) questionnaires from baseline to 24, 36, 48 and 72 weeks.
  Impact of Events Scale Revised (IES-R)
  22 item patient reported outcome to measure affect of routine life stress, everyday traumas and acute stress, and potential Post Traumatic Stress Disorder (PTSD). Each question is answered from 0 to 4.
  0- Not at all
  1. A little bit
  2. Moderately
  3. Quite a bit
  4. Extremely
  Scores 24 or higher- PTSD is a clinical concern Scores 33 or higher- best cutoff for probable diagnosis of PTSD Scores 37 or higher- enough to suppress immune system
Changes from baseline and evidence of disease progression per the Quality of Life reported outcomes- PROMIS-29 + 2 Profile | 72 weeks
  Change from baseline Quality of Life (QoL) questionnaires from baseline to 24, 36, 48 and 72 weeks.
  PROMIS-29 + 2 Profile
  31- item patient reported outcome to measure physical function, anxiety, depression, fatigue, sleep disturbance, social roles, cognition, and pain in adults.
Examine the effects of COVID-19 on the presence of molecular biomarkers associated with Interstitial Lung Disease | 72 weeks
  Biomarkers prognostic for progression in PF patients incl. Soluble intercellular adhesion molecule-1 (sICAM-1), Surfactant protein D (SP-D), cancer antigen 125 (CA-125), cancer antigen (CA19-9), matrix metalloproteinase7 (MMP7), Krebs von den Lungen-6 (KL-6)
  Biomarkers elevated in PF (vs age-matched controls) incl. cancer antigen 125 (CA-125), Carbohydrate antigen 19-9 (CA19-9), Krebs von den Lungen-6 (KL-6), Surfactant protein D (SP-D), C-C Motif Chemokine Ligand 18 (CCL18), matrix metalloproteinase7 (MMP7), von Willebrand factor (vWF)
  Biomarkers elevated in COVID-19 patients incl. ferritin, Interleukin 6 (IL-6), C-reactive protein (CRP) , monocyte chemoattractant protein-1 (MCP1), Macrophage Inflammatory Protein-1 alpha (MIP1a), Vascular endothelial growth factor (VEGF), basic fibroblast growth factor (bFGF), platelet derived growth factor (PDGF)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Kaner, MD, Principal Investigator — WCM Associate Professor of Clinical Medicine Associate Attending; Craig S Conoscenti, MD, Principal Investigator — Boehringer Ingelheim; Nina Patel, MD, Principal Investigator — Boehringer Ingelheim
Locations (4):
- United States (4):
  - Washington University of St. Louis, St Louis, Missouri
  - New York University Langone Medical Center, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided